CLINICAL TRIAL: NCT06912581
Title: Management of Virgin Abdomen SBO With a 2-year Follow-up
Brief Title: Small Bowel Obstruction in Virgin Abdomen
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Collaborators: North Estonia Regional Hospital (Unknown)
Responsible Party: Principal Investigator, Liis Jaanimäe, General surgeon, PhD student, University of Tartu
Other Study IDs: 377/T-6
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Small Bowel Obstruction Adhesion
Keywords: virgin abdomen SBO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective study conductet at Estonia's two regional hospitals. The data of patients hospitalised for SBO (small bowel obstruction) between 2015-2019 is retrospectively analysed. All other patients are excluded- except for previously unoperated ones (virgin abdomen). Study group analyses whether patients were operated on or was conservative management initiated. It will be studied, if any further medical studies have been done within 2 years of hospitalisation.

DETAILED DESCRIPTION:
Background: The surgical dogma of mandatory operative management of small bowel obstruction (SBO) in patients without prior abdominal operations was re-evaluated by the World Society of Emergency Surgery (WSES) in 2021. A few publications exist on this topic, with a modest number of patients included. The purpose of this study was to analyze the causes and management of small bowel obstruction (SBO) in patients without prior abdominal surgeries.

Methods: Study group retrospectively examined the data of patients hospitalized with SBO from 2015 to 2019. Patients without previous abdominal surgeries-virgin abdomen (VA) were included. Eligible patients' data was evaluated. It was noted whether surgery was performed or conservative management was initiated. In the latter case, information about radiological or endoscopic studies, hospitalizations, or surgeries performed within 2 years after the primary hospitalization was extracted

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with SBO Have not been operated previously

Exclusion Criteria:

Age less than 18 years History of previous operatsions Large bowel obstruction Dynamic ileus

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised for SBO
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
SBO resolution at admission | within hospitalisation
  Patients who have been admitted. The primary outcome measure is SBO resolution within hospitalisation. Usually the conservative treatment is safe and feasible if no alarming symptoms (suggesting bowel ischaemia) are present (but can be prolonged op to 120 hours). Guidelines suggest conservative management up to 72 hours, but no clear guideline is present.
  The resolution will be assessed clinically- return of bowel movement and passing of gas or radiologically- CM in the large bowel in the follow-through.

CONTACTS AND LOCATIONS:
Locations (1):
- Tartu univeristy clinic, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Yes
All data generated or analyzed during this study are included in this article. Further enquiries can be directed to the corresponding author.